CLINICAL TRIAL: NCT04785183
Title: Early Supplementation of Melatonin in Preterm Newborns: the Effects on Oxidative Stress
Brief Title: Antioxidant Effects of Melatonin in Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42/18 - 2018
Record Dates: First submitted 2021-02-16; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Newborn Morbidity; Oxidative Stress; Pre-Term; Melatonin Deficiency
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin Group (Experimental)
  Interventions: Dietary Supplement: Melatonin drops
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin drops — Melatonin oral administration
  Arms: Melatonin Group
Other: Placebo — Oral 5% glucose
  Arms: Control Group

SUMMARY:
Preterm infants are at risk of free radical mediated diseases from oxidative stress (OS) injury. Melatonin (MEL) is a powerful antioxidant and scavenger of free radicals. In preterm neonates, melatonin deficiency has been reported. Several studies tested the efficacy of melatonin to counteract oxidative damage in diseases of newborns such as chronic lung disease, perinatal brain injury, necrotizing enterocolitis, retinopathy of prematurity and sepsis, giving promising results. In these studies, the dosages of melatonin varied over a wide range. The present study was designed to test the hypothesis that oral administration of melatonin reduced OS and consequentially, the occurrence of intraventricular haemorrhage (IVH), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP) and bronchopulmonary dysplasia (BPD) in preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <37 weeks
* Normal liver function tests
* Normal kidney function tests

Exclusion Criteria:

* All babies not born in the clinic
* All babies with severe congenital malformations
* Sepsis
* Inborn errors of metabolism
* Babies suffering from perinatal asphyxia
* Babies born from mothers with mental disorders
* Sample hemolysis
* Insufficient sample
* withdraw informed consent.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Measurement of the melatonin concentration | All participants will be evaluated at 24 hours of life
  Analysis of melatonin concentration in treated group (MEL group) and controls (placebo group)
Measurement of the melatonin concentration | All participants will be evaluated at 48 hours of life
  Analysis of melatonin concentration in treated group (MEL group) and controls (placebo group)

SECONDARY OUTCOMES:
Measurement of AOPP | All participants will be evaluated at 24 hours of life
  Evaluation of advanced oxidative protein products (AOPP) in treated group (MEL group) and controls (placebo group)
Measurement of NPBI | All participants will be evaluated at 24 hours of life
  Evaluation of non protein binding iron (NPBI) in treated group (MEL group) and controls (placebo group)
Measurement of isoprostanes | All participants will be evaluated at 24 hours of life
  Evaluation of isoprostanes in treated group (MEL group) and controls (placebo group)
Measurement of AOPP | All participants will be evaluated at 48 hours of life
  Evaluation of advanced oxidative protein products (AOPP) in treated group (MEL group) and controls (placebo group)
Measurement of NPBI | All participants will be evaluated at 48 hours of life
  Evaluation of non protein binding iron (NPBI) in treated group (MEL group) and controls (placebo group)
Measurement of isoprostanes | All participants will be evaluated at 48 hours of life
  Evaluation of isoprostanes in treated group (MEL group) and controls (placebo group)

OTHER OUTCOMES:
Evaluation of the free radical diseases of prematurity occurence | At 3 months of life
  Evaluation of the occurrence of intraventricular haemorrhage (IVH), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP) and bronchopulmonary dysplasia (BPD)

CONTACTS AND LOCATIONS:
Locations (1):
- Eloisa Gitto, Messina, Italy